CLINICAL TRIAL: NCT01302314
Title: Cognitive Rehabilitation in Patients With Spina Bifida: Effects on Executive Functions, Psychological and Health Related Factors
Brief Title: Cognitive Rehabilitation in Patients With Spina Bifida
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jan Stubberud (Other)
Collaborators: University of Oslo (Other); NYU Langone Health (Other); The Rusk Institute of Rehabilitation Medicine (Unknown); Rotman Research Institute at Baycrest (Other); University of Toronto (Other)
Responsible Party: Sponsor-Investigator, Jan Stubberud, Neuropsychologist and PhD student, Sunnaas Rehabilitation Hospital
Organization: Sunnaas Rehabilitation Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSØ-2011041
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Executive Dysfunction; Cognitive Deficits; Spina Bifida
MeSH Terms: conditions — Cognition Disorders; Spinal Dysraphism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cognitive rehabilitation (Experimental)
  Interventions: Behavioral: Goal management training (GMT)

INTERVENTIONS:
Behavioral: Goal management training (GMT) — Fourteen hours of GMT during a time period of three months.

SUMMARY:
This study will examine the effects of a theoretically grounded and manualized cognitive rehabilitation program on patients with Spina Bifida (SB). SB is often associated with deficit in higher order control over cognition, emotion and behaviour; which is typically referred to as executive functions. The present study will examine the efficacy of Goal Management Training (GMT) in patients with SB that experience executive difficulties. It is expected that GMT will have a favourable effect on cognitive executive functioning, psychological and health related factors.

DETAILED DESCRIPTION:
INTRODUCTION:

Rationale and purpose:

Rehabilitation of impaired cognitive processes has come to be a standard component of medical care after traumatic brain injury (TBI) or stroke (Cicerone, Dahlberg, Malec, Langenbahn, Felicitti, Kneipp, et al., 2005), and sometimes for patients with infections of the brain, hypoxic brain damage, and progressive conditions (Wilson, 2008).

The objective of this study is to determine the effects of a recently developed cognitive rehabilitation program; Goal Management Training (GMT) on the executive functioning in people with SB that have cognitive complaints. To date, research efforts have only focused on categorizing cognitive impairments in SB with no research directed towards rehabilitation for these impairments. Given the extent, nature, and ramifications of cognitive impairments in SB, studies on compensatory-based cognitive rehabilitation that teaches management strategies such as GMT may be beneficial for this population. The research questions in this study are (1) What effect does GMT have on cognitive executive functions? Furthermore, what effect does GMT have on subjective and informant evaluation of executive functioning? (2) What effect does GMT have on mental health and quality of life? (3) What effect does GMT have on coping strategies? There will be a 6 months follow-up with regard to the research questions. It is expected that GMT will have a favourable effect on executive functioning, psychological and health related factors in patients with SB.

BACKGROUND:

Medical and cognitive aspects in Spina bifida (SB):

SB is a birth defect caused by incomplete neural tube development, resulting in a protrusion of spinal cord, meninges, and nerve roots through an opening in the spine. SB is a disorder associated with a variety of brain abnormalities, usually including a congenital malformation of the cerebellum and hindbrain (Chiari II) and in about half the cases, partial dysgenesis of the corpus callosum (Barkovich, 2000). Hydrocephalus occurs in 95% of children with this disorder, with 80-90% requiring shunting (Fletcher et al., 2005). SB represents a complicated series of neural insults that begins prior to birth, with persisting effects on development, including problems in the orthopaedic, cognitive, and behavioural domains (Barkovich, 2000; Dicianno, Kurowski, Yang, et al., 2008).

Executive dysfunction:

Executive functions are higher level cognitive operations involved in the control and direction of lower level functions. Patients with executive dysfunction may experience, problems in dealing with novel situations, problems forming a reasonable plan that takes into account the relevant details, problems inhibiting habitual responses to situations when these are inappropriate, increased distractibility, problems in sustaining attention to task over time and keeping goals on-line, impaired monitoring and error-correction of behavioural output, low motivation, lack of foresight regarding the effects of one's behaviour, difficulty in regulating emotional state, and poor insight into one's difficulties (Levine, Stuss, Winocur, Binns, et al., 2007). Executive dysfunction will be examined in the present study because of the major implications deficits in this cognitive domain have for patients.

Although executive dysfunction is often associated with frontal lobe damage, it can also result from damage to other brain areas. Damage to the frontal-subcortical white matter circuits, which commonly occurs in SB, can disrupt communication between the prefrontal cortex and other areas of the brain (Dennis et al., 2006).

Cognitive rehabilitation:

Cognitive rehabilitation can be defined as a process whereby people with brain injury work together with professional staff and others to remediate or alleviate cognitive deficits arising from a neurological insult (Wilson, 2008). Treatment goals may vary, but the major goal of cognitive rehabilitation is to enable people with disabilities to function as adequately as possible in their own environments (Wilson, 2008). The effectiveness of cognitive rehabilitation is well documented within some domains for patients with stroke and TBI (e.g., Cicerone et al., 2000, 2005; Wilson, 2008; Rees et al., 2007).

The cognitive domain in focus of the present study will be executive functioning. Interventions within this domain, such as Goal Management Training (GMT), include those explicitly directed towards bridging the gap between intention and action, a deficit described as "goal neglect" with interventions targeted towards re-establishing endogenous control of behaviour.

Goal Management Training (GMT):

The present study has translated, and will use an intervention protocol that was originally developed to teach patients with brain injury a strategy to improve their ability to plan activities and to structure intentions; GMT. GMT aims to increase participants' understanding of their own goal management problems, to give them a vocabulary to describe the problems, and to give them a set of techniques to compensate for them.

GMT has been evaluated in 30 patients with mild to severe brain injury, who were randomly assigned to groups who received GMT or motor skill training. Participants who followed the GMT showed significant gains on everyday paper-and-pencil tasks designed to mimic tasks that are problematic for patients with deficits in executive functioning (Levine, Robertson, Clare, Carter, Hong, & Wilson, et al., 2000). Furthermore, Levine et al. (2007) have also applied a version of this protocol in a sample of 49 elderly with subjective cognitive complaints where results indicated improvements in simulated real-life tasks and self-rated executive deficits. These gains where maintained at long-term follow-up. Moreover, in a Dutch study (van Hooren et al., 2007) involving 37 older adults with executive difficulties, the participants in the intervention group were significantly less annoyed by their cognitive failures, were better able to manage their executive failures and reported less anxiety symptoms than those in the waiting list control group after receiving GMT.

METHODS:

The study is an experimental repeated measures design with one treatment group (n=24) and one control group (n=14), total (n=38).

Procedure:

All the patients between the age of 20 and 45 registered at TRS national resource centre for rare disorders in Norway have been asked to participate in the study (n=201). Along with the invitation was a self-report questionnaire, Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A), which the respondents had to fill out and return. Inclusion of patients was based upon one or more elevated scales on the Metacognition Index (MI). Fifty-three (n=53) subjects responded and returned the BRIEF-A questionnaire, and all fulfilled the inclusion criteria.

The baseline measurement of fifty-three (n=53) subjects in this randomised controlled trial (RCT) have been done. At baseline the participants filled out questionnaires concerning cognitive functioning, mental health, quality of life, and coping. Furthermore, neuropsychological assessments were conducted. Additionally, the Dysexecutive Questionnaire and BRIEF-A informant report form were filled out by an adult informant who were familiar with the rated individual's everyday functioning. Six subjects were excluded at baseline because they met the exclusion criteria, six subjects met the inclusion criteria but could not follow the programme at the time being because of hospitalization/illness, and three subjects could not follow the programme at the time being because of school/education. After the baseline measurement the participants were randomly assigned to GMT or control group (waiting list). The method of randomisation was a block design with block size 2, with stratification for age and education.

Twenty-four (n=24) subjects have been assigned to GMT, with six subjects in each GMT training group. The GMT is structured into seven modules. Each module is designed to run for approximately two hours. As such, the subjects will stay at TRS for three days and go through module 1 and 2. Then they go home for a month, come back and stay for three days while going through modules 3, 4 and 5. Once more, they go home for a month, come in and go through modules 6 and 7. GMT consists of tasks performed during training designed to illustrate goal management concepts in action, and homework assignments designed to facilitate transfer of the concepts to real life. Both the control group and the intervention group will be assessed immediately after the intervention group has completed the intervention, and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Spina bifida with myelomeningocele (MMC)
* Between 20 and 46 years of age
* Problems in the domain of executive functioning

Exclusion Criteria:

* Major psychiatric disorder
* Reported alcohol or substance abuse within the past year
* Aphasia or other specified language problems causing potential validity problems
* IQ < 70

Ages: 20 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Self and informant report of cognitive difficulties | Baseline, 3 months and 6 months
  Behavior Rating Inventory for Executive Functions (BRIEF-A; Gioia et al., 2000).
Self and informant report of cognitive difficulties | Baseline, 3 months, and 6 months
  The Dysexecutive Questionnaire (DEX; Burgess, Alderman, Emslie, Evans & Wilson, 1996).
self report of cognitive failures | baseline, 3 months, and 6 months
  Cognitive Failures Questionnaire (Broadbent, Cooper, FitzGerald, & Parkes, 1982).
self report of psychological problems | baseline, 3 months, and 6 months
  Symptom Checklist 25 (SCL-25; Derogatis, 1994).
self report of quality of life | baseline, 3 months, and 6 months
  SF36 (Ware & Sherbourne, 1992).
Self report of coping strategies | baseline, 3 months, and 6 months
  General Coping Questionnaire (GCQ-30; Joseph, Williams & Yule, 1992a).

SECONDARY OUTCOMES:
Cognitive functions measured by neuropsychological tests | Baseline, 3 months and 6 months
  Tower from Delis- Kaplan Executive Function System (D-KEFS; Delis, Kaplan & Kramer, 2001).
Cognitive functions measured by neuropsychological tests | baseline, 3 months and 6 months
  TMT from Delis- Kaplan Executive Function System (D-KEFS; Delis, Kaplan & Kramer, 2001).
Cognitive functions measured by neuropsychological tests | baseline, 3 months, and 6 months
  Stroop from Delis- Kaplan Executive Function System (D-KEFS; Delis, Kaplan & Kramer, 2001).
Cognitive functions measured by neuropsychological tests | baseline, 3 months and 6 months
  Conners Continuous Performance Test II (CPT-II; Conners, 2000)
Cognitive functions measured by neuropsychological tests | baseline, 3 months and 6 months
  The Hotel Task (Manly, Hawkins, Evans, Woldt, & Robertson, 2002).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Stubberud, Psychologist, Principal Investigator — Sunnaas Rehabilitation Hospital
Locations (1):
- Sunnaas rehabilitation hospital, Oslo, Nesoddtangen, Norway